CLINICAL TRIAL: NCT03166449
Title: Effects of Immunonutrition on Biomarkers in Traumatic Brain Injury Patients in Malaysia: a Prospective Randomized Controlled Trial.
Brief Title: Effects of Immunonutrition on Biomarkers in Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Loh Pui San, Consultant Anesthesiologist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-1430-23171.
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Traumatic Brain Injury; Immuno-Deficiency; Nutrient Deficiency
Keywords: Traumatic Brain injury; Immunonutrition
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neomune (Experimental): 18 patients with traumatic brain injury were given Neomune as enteral nutrition.
  Interventions: Dietary Supplement: Neomune
- Fresubin® HP energy (Active Comparator): 18 patients with traumatic brain injury were given Fresubin® HP energy as enteral nutrition.
  Interventions: Dietary Supplement: Fresubin® HP energy

INTERVENTIONS:
Dietary Supplement: Neomune — Enteral feeding with Neomune was delivered within 24 to 48 h after admission or surgery according to Brain Trauma Foundation (BTF) Guidelines
  Arms: Neomune
Dietary Supplement: Fresubin® HP energy — Enteral feeding with Neomune was delivered within 24 to 48 h after admission or surgery according to Brain Trauma Foundation (BTF) Guidelines
  Arms: Fresubin® HP energy

SUMMARY:
Background: Head injury is one of the top three diagnosis leading to intensive care unit (ICU) admission in Malaysia. There has been growing interest in using immunonutrition as a mode of modulating the inflammatory response to injury or infection with the aim of improving clinical outcome. The aim of the present study was to evaluate the effect of an immunonutrition on biomarkers (IL-6, glutathione, CRP, total protein and albumin) in traumatic brain injury patients.

Methods: Thirty six patients with head injury admitted to neurosurgical ICU in University Malaya Medical Centre were recruited for this study, over a 6-month period from July 2014 to January 2015. Patients were randomized to receive either an immunonutrition (Group A) or a standard (Group B) enteral feed. Levels of biomarkers were measured at day 1, 5 and 7 of enteral feeding.

Results: Patients in Group A showed significant reduction of IL-6 at day 5 (p<0.001) with concurrent rise in glutathione levels (p= 0.049). Patients in Group A also demonstrated a significant increase of total protein level at the end of the study (day 7).

Conclusion: These findings indicate the potential of immunonutrition reducing cytokines and increasing antioxidant indices in patients with TBI. However, further studies incorporating patient outcomes are needed to determine its overall clinical benefits.

DETAILED DESCRIPTION:
Introduction:

In 2014, injury ranked fifth as the most common cause of hospitalisation in Malaysia, with 86% of major trauma patients sustaining injuries to head and neck. It is known that injuries to the brain is among the most likely to result in death and disability. Therefore, it was unsurprising when the Malaysian Registry of Intensive Care reported head injury as one of the top three diagnosis leading to intensive care unit (ICU) admissions with an in-hospital mortality rate of 22.1%. In addition to causing a significant problem in Malaysia, injury related mortality and morbidity also affects countries worldwide and is expected to be a major cause of death and disability by the year 2030.

This study aims to evaluate the effect of a specific immunonutrition, Neomune, on biomarkers (cytokines, acute phase serum proteins and antioxidants) in traumatic brain injury patients. This immune enhancing enteral feed contains arginine, glutamine and omega-3 fatty acid.

Methods:

This study and its protocol was approved by the Medical Ethics Committee University Malaya Medical Center (MEC ID NO: 20143-15). Written informed consent was obtained from patient's next of kin.

A prospective randomized controlled trial in patients with head injury comparing two high energy protein enteral formula; Neomune (manufactured by Thai Otsuka Pharmaceutical Co., Ltd., Thailand) and Fresubin® HP (manufactured by Fresenius Kabi, Bod Hamburg, Germany) was conducted. Fresubin® HP energy is the standard enteral feeding used in neurosurgical ICU patients in University Malaya Medical Centre. Neomune was chosen to study its immune-modulating effects.

Patients receiving Neomune were classified as Group A (n=18), whereas those receiving Fresubin® HP energy as Group B (n=18). Neomune is enriched with arginine, glutamine and omega-3 fatty acid.

Subject recruitment criteria:

Thirty six patients with head injury admitted to neurosurgical ICU, University Malaya Medical Centre were recruited for this study, over a 6-month period from July 2014 to January 2015. Patient's inclusion criteria were a) age between 15-78 years old, b) admission within 48 hours of post traumatic event, c) moderate to severe head injury (Glasgow Coma Scale 3-12) and, d) requiring enteral nutrition. Exclusion criteria were a) history of uncontrolled diabetes mellitus, b) history of renal or liver dysfunction, c) severe sepsis with multi organ failure and d) history of significant abdominal or chest injuries requiring major surgery.

Feeding protocol:

Eligible patients were randomized into receiving either Neomune (Group A) or Fresubin® HP energy (Group B) using a computerized random number generator. Fresubin® HP energy is a premixed formula with an energy of 1.5kcal/ml. Neomune formula comes in powder form and thus was prepared to reach a concentration of 1.5kcal/ml in order to make it comparable for the trial.

Enteral feeding was delivered within 24 to 48 h after admission or surgery according to Brain Trauma Foundation (BTF) Guidelines [6]. All feeding were introduced via nasogastric tube and carried out using infusion pump. Enteral feeding was commenced at an initial rate of 20 ml/h, and increased by 20 ml/h every 6 hours until target calorie was reached, provided that there was no significant gastric residual volume (<300 mL). The target calorie for each patient was determined by the clinician working alongside the dietitian using Harris Benedict equation which measures Resting Energy Expenditure (REE). This was further corrected 140% of REE based on studies done on traumatic brain injured patients and nutrition guidelines published by the BTF, the American Association of Neurological Surgeons, and the Joint Section on Neurotrauma and Critical Care. Patients going for scheduled surgery are kept nil by mouth 6 hours prior surgery. Feeding interruption are also kept to a minimal if patients are undergoing procedures, extubation or imaging.

Data collection:

Venous blood was withdrawn from patients at day 1, 5 and 7 of enteral nutrition to measure the levels of interleukin-6 (IL-6), glutathione, C-reactive protein (CRP), total protein and albumin. The concentration of IL-6 and glutathione were determined by ELISA (R&D Systems, Minneapolis, USA) according to manufacturer's protocol. Prealbumin was not included as a nutritional biomarker in this study because this test is not available in our standard laboratory test. Furthermore, we were also limited by resource constraint. All measured outcomes were compared between Group A and Group B.

Sample size analysis:

The sample size for this study was calculated based on a similar study done previously on immune enhancing nutrition in traumatic brain injury by Painter et al.

Statistical analysis The data were analysed using SPSS (Statistical Package for the Social Sciences) software version 20.0. Paired t-test was used to compare the concentration of cytokines, acute phase serum proteins and antioxidants between day 1, 5 and 7 after the administration of enteral feeding. Independent sample t-test was used to compare continuous data which include cytokines, acute phase serum proteins and antioxidant levels between Group A and Group B. Statistical significance was predetermined at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Admission within 48 hours of post traumatic event
* Moderate to severe head injury (Glasgow Coma Scale 3-12)
* Requires enteral nutrition.

Exclusion Criteria:

* Uncontrolled diabetes mellitus
* Renal or liver dysfunction
* Severe sepsis with multi organ failure
* History of significant abdominal or chest injuries requiring major surgery.

Ages: 15 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Levels of biomarkers | Day 1 of enteral nutrition
  Venous blood was withdrawn from patients to check levels of interleukin-6 (IL-6), glutathione, C-reactive protein (CRP)
Levels of biomarkers | Day 5 of enteral nutirtion
  Venous blood was withdrawn from patients to check levels of interleukin-6 (IL-6), glutathione, C-reactive protein (CRP)
Levels of biomarkers | Day 7 of enteral nutirtion
  Venous blood was withdrawn from patients to check levels of interleukin-6 (IL-6), glutathione, C-reactive protein (CRP)

SECONDARY OUTCOMES:
Levels of total protein and albumin | Day 1, 5 and 7 of enteral nutrition
  Venous blood was withdrawn from patients to check levels of total protein and albumin

CONTACTS AND LOCATIONS:
Overall Officials: Vineya Rai Hakumat Rai, Study Chair — University of Malaya
Locations (1):
- Anaesthesia Department, Faculty of Medicine, University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. MOH: National trauma database January 2009 to December 2009 fourth report. 2011. 2. Health Facts 2015 [http://vlib.moh. gov.my/cms/ documentstorage/ com.tms.cms. document.Document_ef876440-a0188549-82a26f00 e6a36876/ KKM_ HEALTH _ FACTS _ 2015.pdf] 3. Hyder AA, Wunderlich CA, Puvanachandra P, Gururaj G, Kobusingye OC: The impact of traumatic brain injuries: a global perspective. NeuroRehabilitation. 2007; 22(5):341-353. 4. MOH: Malaysian registry of intensive care report for 2013. Malaysian Registry of Intensive Care, Clinical Research Centre, Ministry of Health Malaysia; 2013. 5. Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS medicine. 2006;3(11):e442. 6. Bullock MR, Povlishock JT: Guidelines for the management of severe traumatic brain injury. Editor's Commentary. J Neurotrauma. 2007;24 Suppl 1:2 p preceding S1. 7. Harris JA, Benedict FG. A biometric study of human basal metabolism. Proc. Natl. Acad. Sci. 1918;4(12):370-373. 8. Roza AM, Shizgal HM. The Harris Benedict equation reevaluated: resting energy requirements and the body cell mass. Am J Clin Nutr. 1984;40(1):168-182. 9. Painter TJ, Rickerds J, Alban RF. Immune enhancing nutrition in traumatic brain injury-A preliminary study Int J Surg. 2015 Sep 30;21:70-4.
- [Derived] Rai VRH, Phang LF, Sia SF, Amir A, Veerakumaran JS, Kassim MKA, Othman R, Tah PC, Loh PS, Jailani MIO, Ong G. Effects of immunonutrition on biomarkers in traumatic brain injury patients in Malaysia: a prospective randomized controlled trial. BMC Anesthesiol. 2017 Jun 15;17(1):81. doi: 10.1186/s12871-017-0369-4. PMID 28619005